CLINICAL TRIAL: NCT04824274
Title: Transversus Abdominis Plane Block With Intrathecal Fentanyl Versus Intrathecal Morphine in Cesarean Delivery: A Randomized, Controlled, Noninferiority Trial
Brief Title: TAP Block With Intrathecal Fentanyl vs. Intrathecal Morphine in Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-167-1185
Record Dates: First submitted 2021-03-19; First posted 2021-04-01 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Cesarean Section
Keywords: transversus abdominis plane block; morphine; fentanyl; spinal anesthesia; cesarean section; postoperative analgesia
MeSH Terms: interventions — Fentanyl; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus abdominis plane block and intrathecal fentanyl (Experimental): Patients will receive spinal anesthesia with 0.5% bupivacaine 9 mg + fentanyl 10 mcg. Following the completion of surgery, ultrasound-guided bilateral transversus abdominis plane block will be done with 0.375% ropivacaine 15 ml per each side.
  Interventions: Drug: fentanyl; Procedure: Transversus abdominis plane block
- Intrathecal morphine (Active Comparator): Patients will receive spinal anesthesia with 0.5% bupivacaine 9 mg + morphine 75 mcg. Following the completion of surgery, sham block will be done using normal saline.
  Interventions: Drug: morphine; Procedure: Sham block

INTERVENTIONS:
Drug: fentanyl — Fentanyl 10 mcg will be injected intrathecally during spinal anesthesia.
  Arms: Transversus abdominis plane block and intrathecal fentanyl
Drug: morphine — Morphine 75 mcg will be injected intrathecally during spinal anesthesia.
  Other Names: Morphine sulfate
  Arms: Intrathecal morphine
Procedure: Transversus abdominis plane block — Ultrasound-guided bilateral transversus abdominis plane block will be done. 0.375% ropivacaine 15 ml per side will be injected.
  Arms: Transversus abdominis plane block and intrathecal fentanyl
Procedure: Sham block — Ultrasound-guided bilateral transversus abdominis plane sham block will be done. Normal saline 15 ml per side will be injected.
  Arms: Intrathecal morphine

SUMMARY:
This noninferiority study aims to determine whether transversus abdominis plane (TAP) block with intrathecal fentanyl could provide a noninferior analgesia compared with intrathecal morphine after cesarean delivery under spinal anesthesia.

DETAILED DESCRIPTION:
Healthy mothers scheduled to undergo elective cesarean delivery under spinal anesthesia will be randomly allocated to receive either TAP block plus intrathecal fentanyl (Group TF) or intrathecal morphine (Group M).

Primary outcome is pain score with movement at postoperative 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adult full-term parturients scheduled to undergo elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Contraindication to spinal anesthesia
* Any chronic pain unrelated pregnancy
* current opioid medication use
* BMI more than 40 kg m-2
* History of drug allergy or hypersensitivity to fentanyl, morphine, ropivacaine, acetaminophen, NSAIDs, bupivacaine, ramosetron, ondansetron, nalbuphine, Naloxone, metoclopramide
* infection of abdominal wall
* Pregnancy-induced hypertension
* known cardiovascular disease
* Known fetal anomaly
* Any sign of onset of labor

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Pain score with movement at 24 hours after delivery | at 24 hours after delivery
  Pain score with movement at 24hr after delivery, using 11-point Numeric rating scale (0, no pain; 10, the worst pain imaginable)

SECONDARY OUTCOMES:
Intravenous fentanyl consumption | at 6, 12, 18, 24, 48 hours after delivery
  cumulative fentanyl consumption via intravenous patient-controlled analgesia
Pain score at rest | at 6, 12, 18, 24, 48 hours after delivery
  Pain score at rest using 11-point Numeric rating scale (0, no pain; 10, the worst pain imaginable)
Pain score with movement | at 6, 12, 18, 48 hours after delivery
  Pain score with movement using 11-point Numeric rating scale (0, no pain; 10, the worst pain imaginable)
time to first opioid request | during hospital stay, an average of 3 days
  time to first intravenous fentanyl administration from delivery
number of patients requiring rescue analgesics | During the first 48 hour-period after delivery
  number of patients requiring rescue analgesics
Incidence of nausea | During the first 48 hour-period after delivery
  Proportion of patients who experienced nausea
Incidence of vomiting | During the first 48 hour-period after delivery
  Proportion of patients who experienced vomiting
Incidence of pruritus | During the first 48 hour-period after delivery
  Proportion of patients who experienced pruritus
Incidence of sedation | During the first 48 hour-period after delivery
  Proportion of patients who experienced sedation
Incidence of respiratory depression | During the first 48 hour-period after delivery
  Proportion of patients who experienced respiratory depression
Nausea severity | During the first 48 hour-period after delivery
  Nausea severity using 4-point scale with 0=none, 1=mild, 2=moderate, or 3=severe
Pruritus severity | During the first 48 hour-period after delivery
  Pruritus severity using 4-point scale with 0=none, 1=mild, 2=moderate, or 3=severe
Patient satisfaction for overall postoperative managements using 11-point scale (0=totally unsatisfied; 10=totally satisfied) | During the first 48 hour-period after delivery
  Patient satisfaction score for overall postoperative pain managements using 11-point scale (0=totally unsatisfied; 10=totally satisfied)
Hospital length of stay | From admission to hospital discharge, an average of 3 days
  Hospital length of stay (day)
Apgar Score | at 1 minute, at 5 minutes
  Apgar Score of fetus
Umbilical arterial pH | immediately after delivery
  Umbilical arterial pH
Umbilical arterial PO2 | immediately after delivery
  Umbilical arterial PO2
Umbilical arterial PCO2 | immediately after delivery
  Umbilical arterial PCO2

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

REFERENCES:
- [Background] Cole J, Hughey S, Longwell J. Transversus abdominis plane block and intrathecal morphine use in cesarean section: a retrospective review. Reg Anesth Pain Med. 2019 Sep 13:rapm-2019-100483. doi: 10.1136/rapm-2019-100483. Online ahead of print. PMID 31519816
- [Background] Patel SD, Sharawi N, Sultan P. Local anaesthetic techniques for post-caesarean delivery analgesia. Int J Obstet Anesth. 2019 Nov;40:62-77. doi: 10.1016/j.ijoa.2019.06.002. Epub 2019 Jun 8. PMID 31262444
- [Background] Kwikiriza A, Kiwanuka JK, Firth PG, Hoeft MA, Modest VE, Ttendo SS. The analgesic effects of intrathecal morphine in comparison with ultrasound-guided transversus abdominis plane block after caesarean section: a randomised controlled trial at a Ugandan regional referral hospital. Anaesthesia. 2019 Feb;74(2):167-173. doi: 10.1111/anae.14467. Epub 2018 Nov 1. PMID 30383289
- [Derived] Park SK, Kim Y, Kim H, Kim JT. Transversus abdominis plane block combined with intrathecal fentanyl versus intrathecal morphine for post-cesarean analgesia: a randomized non-inferiority clinical trial. Reg Anesth Pain Med. 2025 Jan 21:rapm-2024-106044. doi: 10.1136/rapm-2024-106044. Online ahead of print. PMID 39842942